CLINICAL TRIAL: NCT00220701
Title: Double-Blind Placebo-Controlled Study of Escitalopram in the Treatment of Dysthymic Disorder
Brief Title: Escitalopram in the Treatment of Dysthymic Disorder, Double Blind
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LXP-MD-34
Record Dates: First submitted 2005-09-21; First posted 2005-09-22 (Estimated); Results first posted 2014-11-25 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2007-11

CONDITIONS: Dysthymic Disorder
Keywords: Dysthymic Disorder; Depression; Chronic Depression; Escitalopram
MeSH Terms: conditions — Dysthymic Disorder; Depression | interventions — Escitalopram; Dexetimide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- escitalopram (Experimental): Escitalopram (brand name Lexapro) is an antidepressant medication taken once per day, dosing from 10 to 20 milligrams per day.
  Interventions: Drug: Lexapro (escitalopram)
- Placebo (Placebo Comparator): inactive comparator
  Interventions: Drug: Lexapro (escitalopram)

INTERVENTIONS:
Drug: Lexapro (escitalopram) — antidepressant drug selective serotonin reuptake inhibitor (SSRI)
  Other Names: lexapro; escitalopram; s-citalopram; d-citalopram

SUMMARY:
This is a 12-week double-blind placebo-controlled study of Escitalopram in treatment of dysthymic Disorder (low-grade chronic depression), with a 12 week open-label extension phase.

It is hypothesized that Escitalopram will be superior to placebo in improving depression, as well as psychosocial, temperamental, and cognitive functioning.

DETAILED DESCRIPTION:
This is a 12-week double-blind placebo-controlled study of Escitalopram in treatment of Dysthymic Disorder (low-grade chronic depression), with a 12 week open-label extension phase.

Flexible dosing to a maximum of 40 mg per day will be used. It is hypothesized that Escitalopram will be superior to placebo in improving depression, as well as psychosocial, temperamental, and cognitive functioning. Blood cytokine levels will also be measured at weeks 0, 12, and 24 to determine their relationship to depressive symptoms and improvement.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients 18-65 years of age.
* Patients with a Diagnostic and Statistical Manual, fourth edition (DSM-IV) diagnosis of dysthymic disorder.
* Subject must be considered reliable.
* Patients will have a total of 12 or higher on the Hamilton Depression Scale (24 items) at baseline.

Exclusion Criteria:

* Patients with a DSM-IV diagnosis of Delirium, Dementia, and Amnestic, and other Cognitive Disorders.
* Patients who plan to produce a pregnancy within the next 6 months, or patients who are pregnant or nursing women.
* Patients who have a history of non-response to two or more sufficient trials of antidepressant medication (as defined in Table 1).
* Patients with a principal diagnosis meeting DSM-IV criteria for:

  * Major Depressive Disorder, current
  * Bipolar Disorder or cyclothymia .Schizophrenia, Delusional (Paranoid) Disorders and Psychotic Disorders not elsewhere classified.
  * Anorexia Nervosa or Bulimia
* Patients who, within the past 6 months, met DSM-IV criteria for abuse of or dependence on any drug, including alcohol, excluding caffeine and tobacco.
* Patients who have taken psychotropic medication or herbal preparations with putative psychotropic effects within 7 days prior to Visit 2. Patients taking a monoamine oxidase inhibitor (a type of antidepressant) (MAOI) must have a washout period of 14 days prior to visit 2, and patients taking fluoxetine must have a washout period of at least 4 weeks prior to Visit 2.
* Patients who would pose a serious risk for suicide during the course of the study, as evidenced by one of the following:

  * Report of having a specific plan for killing themselves
  * A score of 3 or higher on the Hamilton Depression Rating Scale item #3 as rated by the treating clinician at Week 0, (indicative of active suicidal thoughts or behaviors)
  * A suicide attempt within the past 12 months requiring emergency room visit, medical or psychiatric hospitalization, or otherwise deemed to be life-threatening (e.g. an overdose of > 1 week's dose of medication.
* Patients with unstable medical conditions, such as acute hyperthyroidism, uncorrected hypothyroidism, undiagnosed fever, uncontrolled angina, or any other serious medical illness, including any cardiovascular, hepatic, respiratory, hematological, endocrinologic o neurologic disease, or any clinically significant laboratory abnormality.
* Patients who lack the capacity to proved informed consent
* 50% or greater decrease in HDRS total score from visit 2 to visit 3 or a CGI-Improvement score of 1 ("very much improved") or 2 ("much improved") at Visit 3
* Patients receiving CGI Improvement scores of 6 ("much worse") or 7 ("very much worse") for two consecutive visits will be withdrawn from the study.
* Patients who meet criteria for Major Depressive Disorder at any time during the course of the study will be withdrawn from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2002-06; Primary Completion 2008-11 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Hellerstein, MD, Principal Investigator — St. Luke's-Roosevelt Hospital, and NY State Psychiatric Institute
Locations (1):
- Mood Disorders Research Program, St. Luke's-Roosevelt Hospital Center, New York, New York, United States

REFERENCES:
- [Result] Hellerstein DJ, Batchelder ST, Hyler S, Arnaout B, Toba C, Benga I, Gangure D. Escitalopram versus placebo in the treatment of dysthymic disorder. Int Clin Psychopharmacol. 2010 May;25(3):143-8. doi: 10.1097/YIC.0b013e328333c35e. PMID 21811192
- See also: For more information about our program and this study click here. — http://www.DepressionNY.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Escitalopram | Placebo
Started | 17 | 17
Completed | 12 | 13
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram | Placebo | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.88 (9.92) | 43.59 (11.33) | 43.74 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 11 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Hamilton-Depression Rating Scale (HDRS-24 Items)
Description: Clinician rated measure of depression, mean score; This study used the 24 item version of the Hamilton Depression Rating Scale; item scores range from 0 to 4 on some items, 0 to 2 or 0 to 3 on other items; range of total score = 0 to 75, with higher score indicating worse depression Response (>50% decrease) Remission (score<=7)
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 17 | 17
units on a scale | 10.88 (5.83) | 16.41 (6.34)
Statistical Analysis 1: Comparison: Escitalopram vs Placebo; Test type: Superiority or Other; p = 0.10, Repeated Measures ANOVA; F statistics = 2.82

2. Secondary Outcome: Clinical Global Impressions - Severity (CGI-S)
Description: Clinician rated severity, score on CGI-S scale ranging from 1 (no pathology) to 7 (extreme pathology)
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 17 | 17
units on a scale | 2.35 (0.93) | 3.41 (1.06)

3. Secondary Outcome: Beck Depression Inventory (BDI)
Description: 21 item patient rated assessment of depression symptoms, with item scores ranging from 0 to 3. Total BDI scores can range from 0 to 63, with higher scores indicating worse depression.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 17 | 17
units on a scale | 15.00 (5.21) | 16.25 (5.12)

4. Primary Outcome: Hamilton-Depression Rating Scale (HDRS-24 Items)
Description: as for outcome 1
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 17 | 17
units on a scale | 22.82 (5.75) | 24.41 (6.25)

5. Secondary Outcome: Clinical Global Impressions - Severity (CGI-S)
Description: Clinician rated severity, score on CGI-S scale ranging from 1 (no pathology) to 7 (extreme pathology)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 17 | 17
units on a scale | 4.06 (0.24) | 4.06 (0.43)

6. Secondary Outcome: Beck Depression Inventory (BDI)
Description: as for outcome 3
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 17 | 17
units on a scale | 6.76 (4.91) | 10.00 (5.16)

ADVERSE EVENTS:
Time Frame: Participants were evaluated weekly for the first two weeks after randomization and then biweekly thereafter till week 12.
Arm/Group | Escitalopram | Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 15/17 | 14/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram (N=17) | Placebo (N=15)
Upset stomach (Gastrointestinal disorders) | 0 (0) | 3 (3)
Decreased Libido (Reproductive system and breast disorders) | 6 (6) | 1 (1)
Delayed Ejection (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Lightheadedness (Nervous system disorders) | 3 (3) | 0 (0)
Other (General disorders) | 3 (3) | 10 (10)

LIMITATIONS AND CAVEATS:
Small double blinded study with limited power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No